CLINICAL TRIAL: NCT05196438
Title: Patterns of Congenital Heart Diseases at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Abdelnaeem Khedewy, resident doctor at pediateric department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-12-05
Record Dates: First submitted 2022-01-03; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collecting statistics about congenital heart patterns and investigations done and interventions done to them — Collecting statistics about congenital heart patterns and investigations done and treatment given or interventions e.g. catheterization or surgical operations done to them

SUMMARY:
Congenital heart diseases (CHD) are structural or functional heart diseases that present at birth even if it is discovered later in life .

Congenital heart disease is caused by disturbance in the normal development of the heart especially during the first 6 weeks of pregnancy. Researchers aren't sure about the exact cause , but they think genetics , certain medical conditions , some medications and environmental factors, such as smoking, may play a role .

CHD in many cases may be asymptomatic and discovered accidently during the routine examination or may be presented by some clinical manifestations (e.g. Cyanosis or Murmers) and /or complications (e.g. Heart Failure Manifestations : Tachycardia , Tachypnea , Dyspnea during feeding , Diaphoresis especially during feeding

,Restlessness, irritability , Hepatomegaly , and Failure To Thrive) .

Recently diagnosis of congenital heart disease is better by using advanced technology e.g. echocardiography, magnetic resonance imaging (MRI), cardiac catheterization, angiography, and radio-active isotopes . and early diagnosis is very important as regard the manangement of the disease .

As medical care and surgical interventions have advanced over time, the treatment of many abnormalities is now available . and many infants and children with congenital heart defects are living longer and healthier lives. Many are living into adulthood, requiring ongoing, lifelong medical care for their conditions .

So information about different aspects of CHD is very important for planning health programs for long-term care and maintenance for these cases .

ELIGIBILITY:
Inclusion Criteria:

* All children from date of birth to age of 12 years old including both genders diagnosed to have CHD .

Exclusion Criteria:

* More than 12 years old .
* Acquired heart diseases
* Children with heart rate abnormalities

Ages: 1 Hour to 12 Years | Sex: All
Age Groups: Child
Study Population: All children from date of birth to age of 12 years old including both genders diagnosed to have CHD .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Patterns of congenital heart disease | one year
  Recording of cases of congenital heart diseases with its patterns or types and recording The Management procedures done to them
Incidence & Prevalence of Patterns of Congenital Heart Diseases in Sohag University Hospital | one year
  Recording Incidence and Prevalence of each Pattern of congenital heart diseases with its types for statistical purposes .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Donofrio MT, Moon-Grady AJ, Hornberger LK, Copel JA, Sklansky MS, Abuhamad A, Cuneo BF, Huhta JC, Jonas RA, Krishnan A, Lacey S, Lee W, Michelfelder EC Sr, Rempel GR, Silverman NH, Spray TL, Strasburger JF, Tworetzky W, Rychik J; American Heart Association Adults With Congenital Heart Disease Joint Committee of the Council on Cardiovascular Disease in the Young and Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Council on Cardiovascular and Stroke Nursing. Diagnosis and treatment of fetal cardiac disease: a scientific statement from the American Heart Association. Circulation. 2014 May 27;129(21):2183-242. doi: 10.1161/01.cir.0000437597.44550.5d. Epub 2014 Apr 24. PMID 24763516
- [Background] Silove ED. Assessment and management of congenital heart disease in the newborn by the district paediatrician. Arch Dis Child Fetal Neonatal Ed. 1994 Jan;70(1):F71-4. doi: 10.1136/fn.70.1.f71. No abstract available. PMID 8117134
- [Background] van der Linde D, Konings EE, Slager MA, Witsenburg M, Helbing WA, Takkenberg JJ, Roos-Hesselink JW. Birth prevalence of congenital heart disease worldwide: a systematic review and meta-analysis. J Am Coll Cardiol. 2011 Nov 15;58(21):2241-7. doi: 10.1016/j.jacc.2011.08.025. PMID 22078432